CLINICAL TRIAL: NCT00000841
Title: A Randomized, Double-Blind, Phase III Study of Indinavir Sulfate With Open-Label Zidovudine (AZT) and Lamivudine (3TC) in Subjects With HIV Infection With CD4 Cell Counts <= 200 Cells/mm3 and >= 6 Months of Prior AZT Experience
Brief Title: A Study of Indinavir Sulfate Plus Zidovudine (AZT) Plus Lamivudine in HIV-Infected Patients Who Have Taken AZT for Six or More Months
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 320; 11294 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Antiviral Agents; Zidovudine; Stavudine; HIV Protease Inhibitors; Lamivudine; Indinavir
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Indinavir; Lamivudine; Stavudine; Zidovudine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine

SUMMARY:
To determine the clinical efficacy of indinavir sulfate or placebo in combination with zidovudine ( AZT ) and lamivudine ( 3TC ) in AIDS patients.

Protease inhibitors such as indinavir sulfate may be effective in patients with advanced HIV disease who have received prior AZT therapy. Since studies suggest that triple drug therapy may have an advantage over both monotherapy and two drug therapy, the combination of indinavir sulfate with AZT and 3TC should be evaluated.

DETAILED DESCRIPTION:
Protease inhibitors such as indinavir sulfate may be effective in patients with advanced HIV disease who have received prior AZT therapy. Since studies suggest that triple drug therapy may have an advantage over both monotherapy and two drug therapy, the combination of indinavir sulfate with AZT and 3TC should be evaluated.

Patients are randomized to receive open-label AZT and 3TC with or without indinavir sulfate for at least 48 weeks. Patients who develop intolerance to AZT or have progressive disease after 24 weeks on study may substitute stavudine ( d4T ) for AZT. Patients are followed at weeks 4, 8, 16, 24, 32, 40, and 48 and every 8 weeks thereafter up to week 96. [AS PER 02/25/97 AMENDMENT: Accrual has been halted because interim analysis has shown triple therapy superior to double-agent therapy. An open label extension phase has been added for the period through 06/30/97. Patients who had been randomized to AZT/3TC are given the option of continuing on assigned ACTG 320 study drugs, crossing over to open-label indinavir, or permanently discontinuing all study therapies and going off study. Patients who were randomized to AZT/3TC plus indinavir or who were crossed to such therapy are given the option of continuing their currently assigned therapies. It is strongly suggested that patients who were on AZT/3TC who wish to receive open-label indinavir consider changing the nucleoside analog component of their regimen if at all possible.] [ AS PER 06/06/97 AMENDMENT: The availability of the current ACTG 320 treatment has been further extended for approximately 12 additional weeks (but not beyond 09/30/97). This extension will allow patients to continue receiving study medications until ACTG 372 is open to accrual (the rollover protocol for subjects originally randomized to the triple drug component of ACTG 320 or who are crossed over due to a confirmed study endpoint is finalized).] [ AS PER 09/15/97 AMENDMENT: Open-label therapy will be provided for no more than 90 days beyond the enrollment of the first subject on ACTG 372.]

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* PCP prophylaxis.

Allowed:

* Topical or oral antifungal agents (other than oral ketoconazole).
* Approved agents for opportunistic infections.
* Antibiotics unless specifically excluded.
* Systemic corticosteroids for no more than 21 days.
* Vitamins.
* Recombinant erythropoietin.
* G-CSF.
* Regularly prescribed medications such as allergy medications, antidepressants, antipyretics, analgesics, oral contraceptives, megestrol, and testosterone.

Concurrent Treatment:

Allowed:

* Acupuncture.
* Visualization techniques.

Patients must have:

* HIV infection.
* CD4 count <= 200 cells/mm3.
* At least 6 months total prior AZT therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Malignancy requiring systemic therapy other than minimal Kaposi's sarcoma.

Concurrent Medication:

Excluded:

* Antiretrovirals other than study drugs.
* Rifabutin and rifampin.
* Investigational drugs other than indinavir sulfate.
* Systemic cytotoxic chemotherapy.
* Oral ketoconazole.
* Chronic systemic corticosteroids.
* Herbal therapies.

Patients with the following prior conditions are excluded:

* Unexplained temperature > 38.5 C for any 7 days within 30 days prior to study entry.
* Chronic diarrhea persisting for 15 days within 30 days prior to study entry.
* History of acute or chronic pancreatitis.
* Acute hepatitis within 30 days prior to study entry.
* Grade 2 or worse bilateral peripheral neuropathy within 60 days prior to study entry.
* Dose-limiting intolerance to prior AZT at 600 mg/day.

Prior Medication:

Excluded:

* More than 1 week of prior 3TC.
* Any prior protease inhibitors.
* Rifampin or rifabutin within 14 days prior to study entry.

Excluded within 30 days prior to study entry:

* Erythropoietin.
* G-CSF or GM-CSF.
* Non-nucleoside reverse transcriptase inhibitors.
* Interferons.
* Interleukins.
* HIV vaccines.
* Any experimental therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1750
Dates: Study Completion 1997-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hammer SM, Study Chair; Squires KE, Study Chair; Fischl MA, Study Chair
Locations (87):
- United States (85):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hosp of Los Angeles, Los Angeles, California
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - San Francisco Gen Hosp, San Francisco, California
  - Stanford at Kaiser / Kaiser Permanente Med Ctr, San Francisco, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Kaiser Permanente Franklin Med Ctr, Denver, Colorado
  - Mountain States Reg Hemo Ctr / Univ of Colorado, Denver, Colorado
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - George Washington Univ / Hershey Med Ctr, Washington D.C., District of Columbia
  - Georgetown Univ Hosp, Washington D.C., District of Columbia
  - Howard Univ, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Emory Univ, Atlanta, Georgia
  - Emory Hemo Comp Evaluation Clinic / East TN Comp Hemo Ctr, Atlanta, Georgia
  - Queens Med Ctr, Honolulu, Hawaii
  - Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Louis A Weiss Memorial Hosp, Chicago, Illinois
  - Illinois Masonic Med Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Univ of Iowa Hosp and Clinic, Iowa City, Iowa
  - Charity Hosp / Tulane Univ Med School, New Orleans, Louisiana
  - Tulane Med Ctr Hosp, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - State of MD Div of Corrections / Johns Hopkins Univ Hosp, Baltimore, Maryland
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Boston Med Ctr, Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Worcester Memorial Hosp / Med Ctr of Cntrl MA-Memorial, Worcester, Massachusetts
  - Hennepin County Med Clinic, Minneapolis, Minnesota
  - Univ of Minnesota, Minneapolis, Minnesota
  - St Paul Ramsey Med Ctr, Saint Paul, Minnesota
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - North Shore Univ Hosp, Great Neck, New York
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Kaplan Cancer Ctr / New York Univ Med Ctr, New York, New York
  - Manhattan Veterans Administration / New York Univ Med Ctr, New York, New York
  - Saint Clare's Hosp and Health Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - St Vincent's Hosp / Mem Sloan-Kettering Cancer Ctr, New York, New York
  - Mount Sinai Med Ctr / Hemophilia Treatment Ctr, New York, New York
  - Mount Sinai Med Ctr / Pediatrics, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - SUNY / State Univ of New York, Syracuse, New York
  - Montefiore Med Ctr Adolescent AIDS Program, The Bronx, New York
  - Bronx Veterans Administration / Mount Sinai Hosp, The Bronx, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Carolinas Med Ctr, Charlotte, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Moses H Cone Memorial Hosp, Greensboro, North Carolina
  - Central Prison/Women's Prison in Raleigh / NC, Raleigh, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Univ of Kentucky Lexington, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - Columbus Children's Hosp, Columbus, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Milton S Hershey Med Ctr, Hershey, Pennsylvania
  - Thomas Jefferson Univ Hosp, Philadelphia, Pennsylvania
  - Med Univ of South Carolina, Charleston, South Carolina
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Tennessee / E Tennessee Comprehensive Hemophilia Ctr, Knoxville, Tennessee
  - Meharry Med College, Nashville, Tennessee
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Univ of Texas Galveston, Galveston, Texas
  - Univ Texas Health Science Ctr / Univ Texas Med School, Houston, Texas
  - Univ of Washington, Seattle, Washington
  - Great Lakes Hemophilia Foundation, Wauwatosa, Wisconsin
- Puerto Rico (2):
  - Ramon Ruiz Arnau Univ Hosp / Pediatrics, Bayamón
  - Univ of Puerto Rico, San Juan

REFERENCES:
- [Background] Reiter G, Wojnarowski C. Low rate of nelfinavir discontinuation in a clinic population. Int Conf AIDS. 1998;12:1049 (abstract no 60273)
- [Background] ACTG 320 trial halted as three-drug arm proves superior. AIDS Patient Care STDS. 1997 Jun;11(3):194. No abstract available. PMID 11361796
- [Background] Conference updates show promising drug data. AIDS Alert. 1997 Nov;12(11):125-6. PMID 11364769
- [Background] Baker R. 3-drug therapy reduces deaths and new AIDS-related illnesses by 50%. BETA. 1997 Mar:3-4. PMID 11364527
- [Background] Demeter LM, Hughes MD, Coombs RW, Jackson JB, Grimes JM, Bosch RJ, Fiscus SA, Spector SA, Squires KE, Fischl MA, Hammer SM. Predictors of virologic and clinical outcomes in HIV-1-infected patients receiving concurrent treatment with indinavir, zidovudine, and lamivudine. AIDS Clinical Trials Group Protocol 320. Ann Intern Med. 2001 Dec 4;135(11):954-64. doi: 10.7326/0003-4819-135-11-200112040-00007. PMID 11730396
- [Background] Demeter LM, Bosch RJ, Coombs RW, Fiscus S, Bremer J, Johnson VA, Erice A, Jackson JB, Spector SA, Squires KM, Fischl MA, Hughes MD, Hammer SM. Detection of replication-competent human immunodeficiency virus type 1 (HIV-1) in cultures from patients with levels of HIV-1 RNA in plasma suppressed to less than 500 or 50 copies per milliliter. J Clin Microbiol. 2002 Jun;40(6):2089-94. doi: 10.1128/JCM.40.6.2089-2094.2002. PMID 12037070
- [Background] Coplan P, Cook J, Carides G, Nguyen BY, Testa M. Impact of indinavir with zidovudine and lamivudine on quality of life for HIV patients with < or = 200 CD4 in ACTG 320. Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:86 (abstract no 101)
- [Background] Hammer SM, Squires KE, Hughes MD, Grimes JM, Demeter LM, Currier JS, Eron JJ Jr, Feinberg JE, Balfour HH Jr, Deyton LR, Chodakewitz JA, Fischl MA. A controlled trial of two nucleoside analogues plus indinavir in persons with human immunodeficiency virus infection and CD4 cell counts of 200 per cubic millimeter or less. AIDS Clinical Trials Group 320 Study Team. N Engl J Med. 1997 Sep 11;337(11):725-33. doi: 10.1056/NEJM199709113371101. PMID 9287227
- [Background] Demeter LM, Degruttola V, Eshleman S, Jackson JB, Hughes M, Hammer SM. Baseline (BL) HIV-1 protease (PR) and reverse transcriptase (RT) genotype as a predictor of response to ZDV+3TC+indinavir (IDV). Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:92 (abstract no 131)
- [Background] Freedberg KA, Goldie SJ, Paltiel AD, Losina E, Cohen CJ, Seage GR, Craven DE, Zhang H, Kimmel AD, Sullivan LM, Weinstein MC. Combination antiretroviral therapy is both effective and cost-effective. 39th Intersci Conf Antimicrob Agents Chemother. 1999 Sept 26-29 (abstract no I-2070)
- [Background] Levine, AM. HPV Infection and Cervical/Anal Precursor Lesions in the HAART Era. http://www.medscape.com/viewarticle/440151
- [Background] Coplan PM, Cook JR, Carides GW, Heyse JF, Wu AW, Hammer SM, Nguyen BY, Meibohm AR, DiNubile MJ; AIDS Clinical Trials Group 320 Study Team. Impact of indinavir on the quality of life in patients with advanced HIV infection treated with zidovudine and lamivudine. Clin Infect Dis. 2004 Aug 1;39(3):426-33. doi: 10.1086/422520. Epub 2004 Jul 19. PMID 15307012
- [Result] Mrus JM, Williams PL, Tsevat J, Cohn SE, Wu AW. Gender differences in health-related quality of life in patients with HIV/AIDS. Qual Life Res. 2005 Mar;14(2):479-91. doi: 10.1007/s11136-004-4693-z. PMID 15892437
- [Result] Mrus JM, Schackman BR, Wu AW, Freedberg KA, Tsevat J, Yi MS, Zackin R. Variations in self-rated health among patients with HIV infection. Qual Life Res. 2006 Apr;15(3):503-14. doi: 10.1007/s11136-005-1946-4. PMID 16547789
- [Result] Cole SR, Stuart EA. Generalizing evidence from randomized clinical trials to target populations: The ACTG 320 trial. Am J Epidemiol. 2010 Jul 1;172(1):107-15. doi: 10.1093/aje/kwq084. Epub 2010 Jun 14. PMID 20547574